CLINICAL TRIAL: NCT02277496
Title: Wellness Program Implementation: School & Student Toolkits
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: HealthCorps (Unknown)
Responsible Party: Principal Investigator, Judith Wylie-Rosett, Assistant Professor, Albert Einstein College of Medicine
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: 2013-2056
Record Dates: First submitted 2014-09-10; First posted 2014-10-29 (Estimated); Last update posted 2018-12-04 (Actual); Status verified 2018-01

CONDITIONS: Overweight; Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Intervention Model Description: During the 2014-2015 school year a 2-arm design was used to compare outcomes between intervention and comparison schools. Subsequent years utilized a single-arm design to analyse trends between and within intervention schools only.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HC toolkit intervention students (Experimental): HC students will receiveeExperimental wellness education via a toolkit approach to address the 2010 Dietary Guidelines for reducing obesity in youth. The specific recommendations include: 1) reducing intake of sugary beverages, 2) increasing intake of fruits and vegetables, 3) increasing frequency of eating breakfast, 4) decreasing fast and junk food choices, 5) increasing physical activity to 1 hour/day, and 6) decreasing screen time to 2 hours per day.
  Interventions: Behavioral: Toolkit Intervention
- Comparison Schools (No Intervention): During the 2014-2015 school year, control schools were utilized to compare outcomes.

INTERVENTIONS:
Behavioral: Toolkit Intervention — The toolkit intervention consists of strategies and activities to engage students (student toolkit) and school wellness councils (school toolkit) in addressing the six targeted behaviors of the 2010 Dietary Guidelines based on the principles of participatory action research. The intervention will promote goal setting and school-based food and physical promotion activities led by students as well as school wellness network development.
  Other Names: Student and School Toolkits
  Arms: HC toolkit intervention students

SUMMARY:
The project is designed to evaluate a participatory implementation model in HealthCorps (HC) high schools and to assess outcomes within and across school settings . The behavioral objectives from the 2010 Dietary Guidelines to address obesity in youth include: 1) decreasing sugary beverage intake; 2) increasing frequency of breakfast; 3) increasing vegetable and fruit intake to 2½ cups per day;4) decreasing frequency of fast food meals;5) becoming physically active (goal of 1 hour per day); and 6) reducing sedentary behavior time (<2 hour day). The study is employing system dynamics modeling (SDM) to assess wellness programming options and to evaluate the program implementation within the context of diverse school ecologies. The RE-AIM evaluation metric (Reach, Effectiveness, Adoption, Implementation, and Maintenance) is used to guide SDM development and validation.

The Specific Aims are:

1. To use PAR (Participatory Action Research) methods to refine the school wellness program model and toolkit components that address institutional/community level program implementation barriers and individual level barriers to achieving healthy lifestyle recommendations.
2. To assess the effectiveness of program components using process evaluation techniques guided by the RE-AIM (Reach, Effectiveness, Adoption, Implementation, and Maintenance) model.
3. To evaluate implementation with system dynamics modeling to facilitate dissemination. The simulation analysis will apply the RE-AIM framework to address: Reach (participation rates), effectiveness (outcomes), adoption (acceptability), implementation (intervention fidelity), and maintenance (sustainability of lifestyle changes by students and programs by schools), in order to facilitate refining the toolkits and training program for dissemination to other school setting and diverse educational venues.

DETAILED DESCRIPTION:
This research project focuses on enhancing implementation of school wellness activities with the goal of achieving federal lifestyle recommendations to reduce obesity. The study will evaluate whether using a toolkit approach with problem-solving and other strategies helps schools and students develop healthier lifestyle choices.

At the school level, we will focus on implementation barriers identified by (or brought to) the school Wellness Champion Network (e.g., crowded gym, lack of equipment, food service issues) using a toolkit approach that builds on the Alliance for a Healthier Generation school toolkits.

At the student level, the toolkit will focus on a self-assessed health-behavior feedback mechanism to personalize behavioral goal setting when addressing obesity related lifestyle recommendations.

An iterative intervention dissemination will be used to achieve sequential roll out to all HealthCorps-affiliated Living Lab schools over time. This design allows for an increasingly larger selection of schools to receive the enhanced support through participation research principles to determine how to address obesity-related school mandates. Consistent with participatory research principles, all HealthCorps coordinators have received training to function as Wellness Council facilitators. This study will evaluate a participatory implementation model designed to extend wellness and stakeholder collaborations towards achieving policy standards and goals focusing on the school wellness network. By the end of the study, all HealthCorps Living Labs schools will be implementing this participatory implementation for wellness programming.

This implementation approach increases the potential for learning lessons that can be generalized more widely as in pragmatic trials. In keeping with participatory research principles, school Wellness Councils will use data obtained during the trial as feedback for potential refinement of their toolkit components.

The research team will work with school Wellness Councils and key stakeholders to develop additional school toolkit items utilizing problem-solving strategies and low-cost methods to address implementation barriers. The elements of participatory action research focus on forming a school Wellness Council partnership to build trust, shared vision, and mutual capacity, and includes engagement at multiple levels as well as active participation of stakeholders to create more salient and effective programs. The HealthCorps coordinator will guide stakeholders via the Wellness Council network and by specific program area to engage in a 6-step iterative process listed below:

1. Examine local indicator data e.g., FitnessGram, Health Behavior Survey with Youth Behavioral Risk Factor Surveillance System (YBRFSS) items, food service data, school environment/climate data, community data
2. Consider how current programs/curricula and alternatives relate to behavioral indicators (using a social ecological framework) to student, family, school, and community consideration of media and other spheres of influence,
3. Develop program/curriculum S.M.A.R.T. (specific, measurable, attainable, realistic and time limited (considering semester/school year)) goals focusing on Dietary Guidelines, mental resilience, and FitnessGram indicators
4. Identify barriers and develop strategies for the school and student toolkit
5. Implement school program elements with ongoing monitoring by stakeholders and the Wellness Council
6. Use an iterative process to adapt to new needs and sustain program

Basic simulation models will be used to demonstrate the potential effects of implementing a given toolkit option. The school and student toolkits developed during the formative evaluation will serve as a template to be used with the intervention schools. The initial training and guide/toolkit formatting will be based on those used by the Alliance for a Healthier Generation in their school wellness programming. Initial feedback from HealthCorps coordinators indicates that the Alliance Wellness Council guide/toolkit can be readily implemented in HealthCorps high schools. The HealthCorps coordinators will build on the Alliance's collaborative guidelines and training to enhance collaboration as an active Wellness Council. In addition, to build youth leadership thereby obtaining student support, the toolkit will include demonstration exercises to be lead by HealthCorps coordinators in collaboration with student leaders and school wellness stakeholders. These demonstration activities, linked to the intervention's behavioral objectives, provide share-able knowledge and skills to promote positive health behavior change.

The outcomes simulation will expand the types of data used to include the survey's psychosocial variables and extensive administrative data such as attendance, demographics, and reduced/free lunch and student, teacher and parent school evaluations.

ELIGIBILITY:
Inclusion Criteria:

* Students (grades 9-12).

Exclusion Criteria:

Ages: 14 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 14520 (Actual)
Dates: Start 2013-07 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Key Behaviors | 12 months
  The primary dependent variables will be the following key behaviors: physical activity, sugary beverage consumptions, fruit and vegetable consumptions and breakfast eating. Scores of these primary study outcomes will be measured annually by administering the high school survey and analyzed cross-sectionally.

SECONDARY OUTCOMES:
Effect of weight changes | 12 months
  The investigators will conduct exploratory analysis to test the effect of weight changes on behavior changes, regardless of intervention assignments. To this end, the investigators will again apply mixed effects linear models in which the dependent variables will be changes in the behavior variables and independent variables will be indicator for direction of changes in BMI z-scores.

OTHER OUTCOMES:
Effects of Goal Setting | 12 months
  Student goal setting behaviors and perceived outcomes will be measured by the research team. This includes the type of goals, the quality of the goals (defined as S-specific, M-measurable, A-actiona oriented, R-realistic, and T-time bound), and the students' perceived success.

CONTACTS AND LOCATIONS:
Overall Officials: Judith Wylie-Rosett, EdD, RD, Principal Investigator — Albert Einstein College of Medicine
Locations (1):
- Albert Einstein College of Medicine, The Bronx, New York, United States

REFERENCES:
- [Derived] Heo M, Jimenez CC, Lim J, Isasi CR, Blank AE, Lounsbury DW, Fredericks L, Bouchard M, Faith MS, Wylie-Rosett J. Effective nationwide school-based participatory extramural program on adolescent body mass index, health knowledge and behaviors. BMC Pediatr. 2018 Jan 16;18(1):7. doi: 10.1186/s12887-017-0975-9. PMID 29338731